CLINICAL TRIAL: NCT05932303
Title: A Phase 1, 3-arm, Open-label, Sequential Design Study to Investigate the Effect of Multiple Doses of Itraconazole, Gemfibrozil, or Carbamazepine on Single-dose Pharmacokinetics of BMS-986278 in Healthy Participants
Brief Title: A Study to Assess the Effect of Multiple Doses of Itraconazole, Gemfibrozil, or Carbamazepine on BMS-986278 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM027-1007
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Healthy Participants
Keywords: BMS-986278; Itraconazole; Gemfibrozil; Carbamazepine; Idiopathic pulmonary fibrosis; Drug interaction
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Itraconazole; Gemfibrozil; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986278, followed by itraconazole (Experimental)
  Interventions: Drug: BMS-986278; Drug: Itraconazole
- BMS-986278, followed by gemfibrozil (Experimental)
  Interventions: Drug: BMS-986278; Drug: Gemfibrozil
- BMS-986278, followed by carbamazepine (Experimental)
  Interventions: Drug: BMS-986278; Drug: Carbamazepine

INTERVENTIONS:
Drug: BMS-986278 — Specified dose on specified days
Drug: Itraconazole — Specified dose on specified days
  Arms: BMS-986278, followed by itraconazole
Drug: Gemfibrozil — Specified dose on specified days
  Arms: BMS-986278, followed by gemfibrozil
Drug: Carbamazepine — Specified dose on specified days
  Arms: BMS-986278, followed by carbamazepine

SUMMARY:
This is a study in healthy participants designed to assess the effect of multiple doses of itraconazole, gemfibrozil, or carbamazepine on the drug levels of a single-dose of BMS-986278.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.0 kilograms per meter squared (kg/m^2) through 32.0 kg/m^2, inclusive.

BMI = weight (kg)/(height [m])2.

* Body weight ≥ 50 kg for males and ≥ 45 kg for females.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Any gastrointestinal disease or surgery (including cholecystectomy) or other procedures (for example, bariatric procedures) that could affect drug absorption, distribution, metabolism, and excretion. Note: Appendectomy is allowed.
* Any major surgery within 4 weeks of study intervention administration.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 33 days
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUC[0-T]) | Up to 33 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 33 days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 33 days
Number of participants with physical examination abnormalities | Up to 33 days
Number of participants with vital sign abnormalities | Up to 33 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 33 days
Number of participants with clinical laboratory abnormalities | Up to 33 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Québec, CA, Canada

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-andresearch/ disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com